CLINICAL TRIAL: NCT01893827
Title: Randomized, Open-label Clinical Trial of Extended-Release vs. Oral Naltrexone for Alcohol Treatment in Primary Care.
Brief Title: Extended-Release vs. Oral Naltrexone Alcohol Treatment in Primary Care
Acronym: X-ON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-02263
Record Dates: First submitted 2013-06-28; First posted 2013-07-09 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Alcohol Dependence
Keywords: Naltrexone; Extended-release naltrexone; Oral naltrexone; Vivitrol; XR-NTX; alcohol dependence; primary care; Medical Management
MeSH Terms: conditions — Alcoholism | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XR-NTX (Active Comparator): Xr-NTX 380mg IM injection monthly x 6 months
  Interventions: Drug: XR-NTX (Extended-Release Naltrexone)
- Oral Naltrexone (Active Comparator): Oral naltrexone 50mg/day x 6 months
  Interventions: Drug: Oral Naltrexone (O-NTX)

INTERVENTIONS:
Drug: XR-NTX (Extended-Release Naltrexone) — 380mg (4cc) XR-NTX administered by IM injection 1x/month for 6 months.
  Other Names: Vivitrol
  Arms: XR-NTX
Drug: Oral Naltrexone (O-NTX) — 50mg pill form of naltrexone taken 1x/day for 6 months.
  Other Names: Revia
  Arms: Oral Naltrexone

SUMMARY:
The proposed study is a pragmatic, randomized, open-label clinical trial of 24 weeks of XR-NTX vs. O-NTX using a COMBINE-adapted Medical Management primary care treatment model. 237 adults >18yo with alcohol dependence will be recruited from the community into treatment in public sector primary care settings. The primary outcome which powers this study is a dichotomous good clinical outcome defined by abstinence or moderate drinking, and as measured by the Timeline Follow-back and analyzed using an intention-to-treat approach among all randomized participants. Secondary outcomes include the incremental cost effectiveness of the two arms, differences between arms by continuous measures of alcohol intake (drinks/day, % days abstinent, time to first heavy drinking day, bio-markers), and the exploratory analysis of factors possibly associated with effectiveness, including gender, prior treatment abstinence, and mu opioid receptor (OPRM1) genotypes.

Specific Aim 1: Treatment Effectiveness. To evaluate the effectiveness of extended-release naltrexone (XR-NTX) vs. oral naltrexone (O-NTX) in producing a primary good clinical outcome, defined as abstinence or moderate drinking (≤2 drinks/day, men; ≤1 drink/day,women; and ≤2 heavy drinking occasions/month), during the final 20 of 24 weeks of primary care-based Medical Management for alcohol dependence. Hypothesis: The rate of this good clinical outcome will be approximately twice as great among participants receiving XR-NTX compared with those receiving O-NTX.

Specific Aim 2: Cost Effectiveness. To estimate the incremental cost effectiveness of XR-NTX vs. O-NTX,both in conjunction with primary care-based Medical Management. Hypothesis: XR-NTX treatment will be more cost effective than O-NTX.

Specific Aim 3: Patient-Level Predictors of Effectiveness. To identify patient-level characteristics associated with effectiveness in both arms.

DETAILED DESCRIPTION:
Rationale: Though integration of alcohol pharmacotherapy into primary care settings is receiving increasing emphasis and support, rigorous data to inform clinicians' treatment choice is lacking. The most recently FDA-approved alcohol treatment medication, an extended-release depot form of naltrexone (XR-NTX, Vivitrol®), could greatly simplify the medical home-centered alcohol treatment emphasized in the National Institute on Alcohol Abuse and Alcoholism (NIAAA) Clinician's Guide. Injected once a month, XR-NTX offers a long-acting and thus potentially more effective form of pharmacotherapy than oral naltrexone (O-NTX), which, despite the Combined Pharmacotherapies and Behavioral Interventions for Alcohol Dependence (COMBINE) trial and systematic reviews supporting some efficacy, has been characterized by low rates of overall prescribing, poor adherence, suboptimal monthly refill and inadequate treatment retention. Yet while promising as an alternative to O-NTX, XR-NTX is substantially more expensive (~$1100 vs. ~$100 per month), and no head-to-head trials have compared the two forms of naltrexone. A comparative effectiveness approach is required to systematically evaluate the following key questions: In primary care settings, what is the relative clinical effectiveness of XR-NTX vs. O-NTX? What are the benefits and costs of XR-NTX relative to O-NTX? And can patient and system characteristics be identified to inform treatment choice to maximize the probability of successful outcome?

Implications: Despite several years of experience, the comparative effectiveness of XR-NTX compared to older alcohol medications remains uncertain, particularly in a mainstream, primary care treatment model that is generalizable and broadly accessible. Newer, novel, expensive medications for addiction disorders are historically greatly underutilized by primary care physicians. This study is innovative both as a 'head-to-head' evaluation of XR-NTX vs. O-NTX in primary care, and because expected participants will be primarily Medicaid-covered or uninsured persons who will not be excluded based on medical and psychiatric co-morbidities that often preclude participation in efficacy studies. If health insurance expansion, parity reforms, medical homes and accountable care organizations are to define primary care as a core alcohol treatment setting in the coming decade, exactly this type of study is required to guide treatment protocols and resource allocation. Ultimately, more widespread adoption of cost-effective alcohol pharmacotherapies will result in longer,healthier lives and lower costs.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age ≥18 y.o.
* English- or Spanish- speaking and able to understand study procedures and provide full consent.
* DSM IV diagnosis of alcohol dependence as determined by study physician and DSM IV checklist.
* Endorses goal of abstinence, and is able to achieve alcohol abstinence without inpatient detoxification, per study physician.

Exclusion Criteria:

* Current opioid dependence and/or positive urine toxicology for extended opioids.
* Pregnancy or female planning conception.
* Allergy to naltrexone or the PGL XR-NTX formulation or diluent.
* Severe liver disease, liver failure, or liver function test levels greater than three times normal.
* Other severe, untreated or uncontrolled medical illness (e.g., severe heart failure or dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D. Lee, MD, MSc, Principal Investigator — NYU School of Medicine, Dept. Population Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | XR-NTX | Oral Naltrexone
Started | 117 | 120
Completed | 98 | 94
Not Completed | 19 | 26
Not completed — Lost to Follow-up | 19 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XR-NTX | Oral Naltrexone | Total
Number analyzed (Participants) | 117 | 120 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (10.6) | 49 (10.7) | 48 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 82 | 84 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 27 | 51
  Not Hispanic or Latino | 93 | 93 | 186
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 67 | 62 | 129
  White | 30 | 44 | 74
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 18 | 12 | 30
Region of Enrollment [Number; unit: participants]
  United States | 117 | 120 | 237

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Alcohol Abstinence or Moderate Drinking
Description: Percentage of participants who had the following number of drinks (≤2 drinks/day, men; ≤1 drink/day, women; and ≤2 heavy drinking occasions/month) during the final 20 of 24 weeks of primary care-based Medical Management for alcohol dependence.
Time Frame: 4-24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | XR-NTX | Oral Naltrexone
Number analyzed (Participants) | 117 | 120
percentage of participants | 29 | 23

2. Other Pre Specified Outcome: Cost-effectiveness
Description: To estimate the incremental cost-effectiveness of XR-NTX vs. O-NTX, both in conjunction with primary care-based medical management. Economic data will be derived primarily from the Economic Form 90, Non-Study Medical Service and electronic medical records assessments, EQ-5D (functional status), and a cost survey or standardized question querying patient reports of specific non-medical related costs (including lost/gained work, lost/gained dependent care, transportation costs, arrests, motor vehicle accidents) collected at baseline and at week 10, 18, 26, and 48 assessments.
Time Frame: 0-24 weeks
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Patient-level Predictors of Effectiveness
Description: To identify patient-level characteristics (gender, ethnicity, pre-treatment abstinence, voluntary specialty alcohol treatment and Alcoholics Anonymous involvement) associated with effectiveness in both arms. Baseline Demographic and Timeline Follow-Back and in-study Non-Study Medical Service questionnaires will characterized these patient-level variables.
Time Frame: 4-24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | XR-NTX | Oral Naltrexone
All-Cause Mortality (participants affected / at risk) | 2/117 | 0/120
Serious Adverse Events (participants affected / at risk) | 22/117 | 20/120
Other Adverse Events (participants affected / at risk) | 19/117 | 18/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XR-NTX (N=117) | Oral Naltrexone (N=120)
Hospitalization (General disorders) | 22 | 20
Death; Stage IV Cancer (General disorders) | 1 | 0
Death; cardiac arrest (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XR-NTX (N=117) | Oral Naltrexone (N=120)
ER Visit (General disorders) | 19 | 18
Scrotal Infection (Infections and infestations) | 1 | 0
Anosmia (General disorders) | 1 | 0
Decreased Libido (General disorders) | 2 | 0
Depressed Mood (Psychiatric disorders) | 1 | 1
Heat Rash (General disorders) | 1 | 0
Hep C (Immune system disorders) | 1 | 0
High Blood Pressure (Blood and lymphatic system disorders) | 1 | 0
HIV (Infections and infestations) | 1 | 0
Nausea (General disorders) | 1 | 0
Nose Fracture (General disorders) | 1 | 0
Rash (General disorders) | 1 | 0
Outpatient Laser Biopsy (Surgical and medical procedures) | 1 | 0
Tooth Extraction (General disorders) | 1 | 0
Cramps (General disorders) | 0 | 1
Dizziness (General disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Insomnia (General disorders) | 0 | 1
Muscle Soreness (General disorders) | 0 | 1
Stomach Pain (General disorders) | 0 | 1
UTI (General disorders) | 0 | 1
Laser Surgery - Outpatient (Surgical and medical procedures) | 0 | 1
CORD/URI (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT01893827/Prot_SAP_000.pdf